CLINICAL TRIAL: NCT00993928
Title: A Randomized Phase II Trial Evaluating Two Non-pharmacologic Interventions in Cancer Survivors for the Treatment of Sleep-wake Disturbances
Brief Title: Home-Based Programs for Improving Sleep in Cancer Survivors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NCCTG-N07C4; NCI-2011-01978 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000656564 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Cancer Survivor; Fatigue; Psychosocial Effects of Cancer and Its Treatment; Sleep Disorders
Keywords: psychosocial effects of cancer and its treatment; fatigue; sleep disorders; cancer survivor
MeSH Terms: conditions — Fatigue; Sleep Wake Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Home-based sleep intervention with Device #1 (Experimental): Participants listen to a pre-recorded mp3 device #1 before retiring to sleep. Only patients in Arm A will have assigned bed and wake times based on their baseline diary.
  Interventions: Behavioral: Home-based sleep intervention
- Arm B: Home-based sleep intervention with Device #2 (Active Comparator): Participants will listen to a pre-recorded mp3 device #2 before retiring to sleep. At the end of the study, participants assigned to pre-recorded mp3 device #2 will be offered pre-recorded mp3 device #1 for their own use.
  Interventions: Behavioral: Home-based sleep intervention

INTERVENTIONS:
Behavioral: Home-based sleep intervention — Participants will be asked to practice behaviors consistent with the stimulus control sheet and to read the sleep hygiene booklet.

SUMMARY:
RATIONALE: Following a program that uses written materials and pre-recorded mp3 devices may help improve the sleep of cancer survivors. It is not yet known which home-based program is more effective in improving the sleep of cancer survivors.

PURPOSE: This randomized phase II trial is comparing two home-based programs for improving sleep in cancer survivors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the efficacy of two home-based sleep interventions as therapy for sleep-wake disturbances,as measured by sleep latency or time to fall back asleep after initial sleep onset per sleep diaries, at baseline (week 1) and at the end of week 7 in cancer survivors.

Secondary

* To compare the efficacy of these interventions as therapy for sleep-wake disturbances as measured by the number of awakenings after sleep, sleep quality, sleep difficulty, and sleep latency at baseline (week 1) and weeks 4 and 7 in these participants.
* To compare the efficacy of these interventions as therapy for sleep-wake disturbances as measured by the percentage of participants in each group who show improved sleep per the Pittsburgh Sleep Quality Index.
* To compare the effects of these interventions on fatigue, mood disturbance, sleep, benefit, and distress in this patient population.
* To describe the side effects associated with these interventions in these patients.
* To describe patient practice habits and adherence measured via a sleep behavior record.
* To explore symptom clusters in this patient population and look at distress as a mediating variable. (Exploratory)
* To explore predictors of sleep quality. (Exploratory)

OUTLINE: This is a multicenter study. Patients are stratified according to current (≥ 1 per week in the past 4 weeks) pharmacological treatment, including anxiolytics, for insomnia or mood (yes vs no), current pharmacologic treatment for pain (yes vs no), sleep difficulty period (≤ 1 month vs > 1 month), and age (≤ 50 vs 51-70 vs > 70 years). Patients are randomized to 1 of 2 intervention groups.

* Group 1: Participants receive a home-based sleep intervention comprising a Sleep Hygiene Education booklet, printed stimulus-control guidelines, instructions on sleeping restrictions, and a guided-imagery pre-recorded mp3 device. Participants meet with study personnel for intervention refinement and are asked to practice behaviors consistent with the stimulus-control sheet, to read the sleep hygiene booklet one chapter per day for 7 days during the first week, and then as needed during study. They are also instructed to use the CD, with or without headphones, in a quiet and comfortable place without lights for up to 30 minutes every day for 6 weeks before bedtime. Participants are instructed to go to sleep and wake at the same time every day during study intervention.
* Group 2: Participants receive a home-based sleep intervention comprising a Sleep Hygiene Education booklet, printed stimulus-control guidelines, and a pre-recorded mp3 device containing short stories and essays. Participants meet with study personnel and are instructed to practice behaviors consistent with the stimulus control sheet, to read the sleep hygiene booklet, and use the CD as in group 1. Participants are not instructed about sleeping restrictions. They are offered the guided-imagery CD after study completion.

Patients complete a Three-Day Sleep Behavior Record for 3 consecutive days at baseline and during weeks 4 and 7 of study intervention. Patients also complete questionnaires on Numeric Analog Sleep for Pain Scale, daily use of CD, Sleep Hygiene Practice, Pittsburgh Sleep Quality Index, Profile of Mood States, Brief Fatigue Inventory, Distress Thermometer, Side-Effect Questionnaire, and a Subject Global Impression of Change at baseline, during weeks 2 and 6, and after completion of study intervention.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Prior diagnosis of cancer
* At least 2 months and ≤ 24 months since completed curative-intent treatment (chemotherapy, surgery, and/or radiotherapy)

  * Ongoing hormonal therapy (i.e., tamoxifen, aromatase inhibitors, casodex)
  * Concurrent trastuzumab and maintenance rituximab allowed
* Sleep difficulty defined as self report of sleep latency of ≥ 30 minutes on 3 out of 7 nights in a week and wishing therapeutic intervention, and/or self report of waking up after first falling asleep and not being able to fall back asleep for ≥ 30 minutes on 3 out of 7 nights in a week
* No history of diagnosis of primary insomnia (patient medical record, defined by having had behavioral, cognitive, or pharmacologic treatment) for > 30 consecutive days in the year before cancer diagnosis
* No active cancer (i.e., not considered no evidence of disease)
* No concurrent CNS malignancy
* No history of diagnosed sleep disorder (i.e., obstructive sleep apnea, restless legs, or periodic leg movement disorder)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Availability of a CD player and head or earphones
* Ability to complete questionnaires
* No uncontrolled chronic pain (i.e., pain score of ≥ 4 on Numeric Analogue Sleep and Pain Scale)
* No diagnosis of major depression disorder, acute anxiety disorder, or schizophrenia per medical record
* No hot flashes that interrupt sleep
* Not working overnight hours and unable to change schedule
* No emotional, psychological, or physical state that, according to physician and/or study personnel evaluation, would preclude adherence to daily home intervention implementation

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 4 days since prior corticosteroid, including inhaled steroids, of any dose for > 2 days
* No prior experience with guided imagery or cognitive behavioral therapy for insomnia
* No concurrent new herbal therapies

  * Stable dose of daily herbal supplements started ≥ 8 weeks before study intervention allowed
  * Herbal teas or herbs in various drink products allowed
* No concurrent treatment with variable doses of any of the following:

  * Antidepressants
  * Anxiolytics
  * Pain medication (not including over the counter ad anti-inflammatory pain relievers)
* Pharmacologic treatment for sleep/wake disturbances is allowed, but must be used for 4 weeks before study entry, and can be used daily or intermittently

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2019-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra Barton, RN, PhD, AOCN, FAAN, Study Chair — Mayo Clinic
Locations (193):
- United States (193):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Lakeland Regional Cancer Center at Lakeland Regional Medical Center, Lakeland, Florida
  - Florida Hospital - Orlando, Orlando, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Oncare Hawaii Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - University of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Oncare Hawaii, Incorporated - Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Weiss Memorial Hospital, Chicago, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Ochsner Clinic Foundation-Baton Rouge, Baton Rouge, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Bixby Medical Center, Adrian, Michigan
  - Toledo Clinic Cancer Centers - Adrian, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Toledo Clinic Cancer Centers - Monroe, Monroe, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Essentia Health - Duluth Clinic, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Central Care Cancer Center-Carrie J Babb Cancer Center, Bolivar, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Mercy-Springfield, Springfield, Missouri
  - Ozark Health Ventures LLC dba Cancer Research for the Ozarks - Springfield, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Cox Medical Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Frontier Cancer Center and Blood Institutes - Billings, Billings, Montana
  - Billings Clinic, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare - Sletten Cancer Institute, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Saint Joseph Hospital, Nashua, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of Central New York PC, East Syracuse, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Toledo Clinic Cancer Centers - Bowling Green, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Health Partners Regional Medical Center - Mercy Cancer Center, Elyria, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Oncology Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers - Oregon, Oregon, Ohio
  - Southern Ohio Medical Center Cancer Center, Portsmouth, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Mercy Cancer Center - Saint Anne Mercy Hospital, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - Greenville Cancer Center of the Carolinas (CCOP), Greenville, South Carolina
  - Cancer Centers of the Carolinas-Greer Medical Oncology, Greer, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Fredericksburg Oncology Inc., Fredericksburg, Virginia
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Gundersen Lutheran Health System/CCOP, La Crosse, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

REFERENCES:
- [Derived] Barton DL, Atherton PJ, Satele DV, Qin R, Dakhil S, Pipe T, Hobday T, Fee-Schroeder K, Loprinzi CL. A randomized phase II trial evaluating two non-pharmacologic interventions in cancer survivors for the treatment of sleep-wake disturbances: NCCTG N07C4 (Alliance). Support Care Cancer. 2020 Dec;28(12):6085-6094. doi: 10.1007/s00520-020-05461-6. Epub 2020 Apr 19. PMID 32307658

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A: Home-based Sleep Intervention With Device #1 | Arm B: Home-based Sleep Intervention With Device #2
Started | 48 | 45
Completed | 43 | 38
Not Completed | 5 | 7
Not completed — Withdrawal by Subject | 4 | 7
Not completed — ineligible | 1 | 0

BASELINE CHARACTERISTICS:
Population: All eligible patients that started protocol treatment were included in baseline analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Home-based Sleep Intervention With Device #1 | Arm B: Home-based Sleep Intervention With Device #2 | Total
Number analyzed (Participants) | 43 | 38 | 81
Age, Continuous [Median (Full Range); unit: years] | 55 [36 to 78] | 59 [31 to 77] | 57 [31 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 32 | 67
  Male | 8 | 6 | 14
Region of Enrollment [Number; unit: participants]
  United States | 43 | 38 | 81

OUTCOME MEASURES:

1. Primary Outcome: Change of the (3 Day) Sleep Latency Time and Time to Fall Back Asleep After Awakening During the Night From Baseline to the End of Study at Week 7
Description: The primary analysis will compare the change in time (in minutes) to fall asleep from baseline to week 7 as reported by question 3 in the sleep diary: "How long did it take you to get to sleep last night?" and time to fall back asleep after awakening during the night as reported by question 6A on sleep dairy: "When waking up after first falling asleep, how long did it take you to fall back to sleep?" >
  > Data were analyzed as a percent change from baseline to week 7. The percent change were compared between arms using a Wilcoxon rank-sum test.
Time Frame: Baseline and 7 weeks
Population: In Arm A, 4 went off treatment prior to week 7 and 2 had missing data. 23 patients were able to respond to question 6A. In Arm B, 7 did not finish 7 weeks of treatment and 1 patient had missing data. 16 patients responded to question 6A. Therefore, Q3 and Q6A are based on 37 and 23 patients in Arm A and 30 and 23 patients from Arm B, respectively.
Measure: Median (Full Range); unit: percentage change
Groups:
- Arm A: Home-based Sleep Intervention With Device #1: Participants listen to a pre-recorded mp3 device #1 before retiring to sleep. Only patients in Arm A will have assigned bed and wake times based on their baseline diary.>
  > Home-based sleep intervention: Participants will be asked to practice behaviors consistent with the stimulus control sheet and to read the sleep hygiene booklet.
- Arm B: Home-based Sleep Intervention With Device #2: Participants will listen to a pre-recorded mp3 device #2 before retiring to sleep. At the end of the study, participants assigned to pre-recorded mp3 device #2 will be offered pre-recorded mp3 device #1 for their own use.>
  > Home-based sleep intervention: Participants will be asked to practice behaviors consistent with the stimulus control sheet and to read the sleep hygiene booklet.
Arm/Group | Arm A: Home-based Sleep Intervention With Device #1 | Arm B: Home-based Sleep Intervention With Device #2
Number analyzed (Participants) | 37 | 30
percentage change
  Q3: Sleep Latency | -25 [-90 to 157] | -45.6 [-90 to 255]
  Q6A: TIme to fall back Asleep: number analyzed (Participants) | 23 | 16
  Q6A: TIme to fall back Asleep | -17 [-91 to 145] | -40 [-86 to 350]
Statistical Analysis 1: Comparison: Arm A: Home-based Sleep Intervention With Device #1 vs Arm B: Home-based Sleep Intervention With Device #2; Comparison of Q3: Percent change in sleep latency from baseline to week 7; Test type: Superiority or Other; p = 0.85, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm A: Home-based Sleep Intervention With Device #1 vs Arm B: Home-based Sleep Intervention With Device #2; Comparison of Q6A: Percent change in time to fall back asleep from baseline to week 7; Test type: Superiority or Other; p = 0.86, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Efficacy of Home-based Interventions on the Number of Awakenings After Sleep, Sleep Quality, Sleep Difficulty, and Sleep Latency at Baseline and Weeks 4 and 7.
Description: Overall efficacy was analyzed as a composite of 4 outcomes: 1. sleep difficulty, 2. sleep quality, 3. Number of awakenings, and 4. Sleep latency. These 4 outcomes were measured by the responses to the following questions, respectively:>
  1. How difficult was it to get to sleep last night? (scale 1-5, 5 meaning very easy)>
  2. How deeply did you sleep last night? (scale 1-5, 5 meaning very deeply)>
  3. How many times did you awaken last night?>
  4. How long did it take you to get to sleep last night?> > The 4 questions were analyzed as percent change from baseline after week 4 and after week 7. The percent change between arms was analyzed using a Wilcoxon test.
Time Frame: Baseline and 7 weeks
Population: In Arm A, 38 patients responded to questions during week 4 and 37 responded during week 7. In Arm B, 31 patients responded during week 4 and 30 responded during week 7.
Measure: Median (Full Range); unit: percentage of change
Arm/Group | Arm A: Home-based Sleep Intervention With Device #1 | Arm B: Home-based Sleep Intervention With Device #2
Number analyzed (Participants) | 43 | 38
percentage of change
  Sleep Difficulty: Week 4: number analyzed (Participants) | 38 | 31
  Sleep Difficulty: Week 4 | 18 [-55 to 200] | 37.5 [-43 to 200]
  Sleep Difficulty: Week 7: number analyzed (Participants) | 37 | 30
  Sleep Difficulty: Week 7 | 20 [-46 to 333] | 45 [-46 to 175]
  Sleep Quality: Week 4: number analyzed (Participants) | 38 | 31
  Sleep Quality: Week 4 | 13 [-25 to 175] | 20 [-30 to 267]
  Sleep Quality: Week 7: number analyzed (Participants) | 37 | 30
  Sleep Quality: Week 7 | 22 [-71 to 200] | 29 [-40 to 233]
  Number of Awakenings: Week 4: number analyzed (Participants) | 38 | 31
  Number of Awakenings: Week 4 | -40 [-100 to 150] | -44 [-100 to 600]
  Number of Awakenings: Week 7: number analyzed (Participants) | 37 | 30
  Number of Awakenings: Week 7 | -50 [-91 to 400] | -48 [-100 to 900]
  Sleep Latency: Week 4: number analyzed (Participants) | 38 | 31
  Sleep Latency: Week 4 | -37 [-83 to 250] | -48 [-92 to 127]
  Sleep Latency: Week 7: number analyzed (Participants) | 37 | 30
  Sleep Latency: Week 7 | -24 [-95 to 700] | -49 [-100 to 91]

3. Secondary Outcome: Comparing the Efficacy of Two Home-based Sleep Interventions as Therapy for Sleep-wake Disturbances as Measured by the Percent of People Who Show Improved Sleep Per the Pittsburgh Sleep Quality Index (PSQI)
Description: The PSQI has 19 items and seven component scales: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep-wake disturbances, use of sleep medication, and daytime dysfunction. The scoring algorithm yields seven component scales on 0-3 scales which are summed to produce a global score on a 0-21 scale with higher values representing more severe sleep difficulty. The percentage of patients that showed improvement or worsening in sleep score from baseline to Week 7 were analyzed and compared using a Chi-squared test.
Time Frame: Baseline and 7 weeks
Population: Thirty-six patients from Arm A and 31 patients from Arm B had PSQI measurements available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Home-based Sleep Intervention With Device #1 | Arm B: Home-based Sleep Intervention With Device #2
Number analyzed (Participants) | 36 | 31
percentage of participants
  Improvement | 36 | 48
  Worsening | 3 | 0
  No Chanage | 61 | 52
Statistical Analysis 1: Comparison: Arm A: Home-based Sleep Intervention With Device #1 vs Arm B: Home-based Sleep Intervention With Device #2; Test type: Superiority or Other; p = 0.42, Chi-squared

4. Secondary Outcome: Total Mood Disturbance as Measured by Profiles of Mood States B (POMS-B)
Description: The POMS-B is a shortened version of the original POMS with 30 items each asking the patient to select how he/she has been feeling during the past week with respect to an adjective such as "tense", "angry", "worn out", etc., on a 0-4 scale (0=not at all; 4=extremely). The POMS-B consists of six identifiable mood states (tension/anxiety, depression/dejection, anger/hostility, vigor/activity, fatigue/inertia, and confusion/bewilderment) and measures the patient's total mood disturbance. This study analyzed total mood disturbance (total scale score) as a secondary endpoints. Possible weekly scores ranged from 0-120. Week 7 scores were analyzed as a percentage change from baseline with a negative score representing a worsening condition. A Wilcoxon rank-sum test was used to compare treatment arms.
Time Frame: At baseline and week 7
Population: Patients that completed the POMS-B questionnaire at baseline and week 7 were used in this analysis.
Measure: Median (Full Range); unit: percentage of change
Arm/Group | Arm A: Home-based Sleep Intervention With Device #1 | Arm B: Home-based Sleep Intervention With Device #2
Number analyzed (Participants) | 34 | 29
percentage of change | 7.8 [-40 to 168] | 7.8 [-15 to 88]

5. Secondary Outcome: Distress at Week 6
Description: The Distress Thermometer is a single-item tool which asks patients to describe how much distress he/she has been experiencing in the past week on a scale of 0 to 10 (0=no distress, 10=extreme distress). The Distress Thermometer was selected for this study due to its brevity. Week 7 distress measures were analyzed as percent change from baseline and analyzed between arms with a t-test.
Time Frame: From baseline to week 7
Population: All patients that completed a Distress Thermometer assessment at baseline and week 7 were included in the analysis.
Measure: Median (Full Range); unit: percentage of change
Arm/Group | Arm A: Home-based Sleep Intervention With Device #1 | Arm B: Home-based Sleep Intervention With Device #2
Number analyzed (Participants) | 35 | 31
percentage of change | 10 [-50 to 70] | 10 [-60 to 70]
Statistical Analysis 1: Comparison: Arm A: Home-based Sleep Intervention With Device #1 vs Arm B: Home-based Sleep Intervention With Device #2; Compare percent change from baseline to week 7 Distress Thermometer score; Test type: Superiority or Other; p = 0.64, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were monitored weekly from week 1 to week 7.
Description: Regardless of whether they completed study treatment or any endpoint, all patients that began intervention and were assessed for adverse events were included in the analysis.
Arm/Group | Arm A: Home-based Sleep Intervention With Device #1 | Arm B: Home-based Sleep Intervention With Device #2
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/43
Serious Adverse Events (participants affected / at risk) | 1/44 | 0/43
Other Adverse Events (participants affected / at risk) | 22/44 | 18/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Home-based Sleep Intervention With Device #1 (N=44) | Arm B: Home-based Sleep Intervention With Device #2 (N=43)
Agitation (Psychiatric disorders) | 1 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Home-based Sleep Intervention With Device #1 (N=44) | Arm B: Home-based Sleep Intervention With Device #2 (N=43)
Facial pain (General disorders) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1)
Periorbital infection (Infections and infestations) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 15 (29) | 10 (22)
Anxiety (Psychiatric disorders) | 19 (49) | 15 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less